CLINICAL TRIAL: NCT04526574
Title: A PHASE 3, RANDOMIZED, DOUBLE-BLIND TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A 20-VALENT PNEUMOCOCCAL CONJUGATE VACCINE (20VPNC) WHEN COADMINISTERED WITH SEASONAL INACTIVATED INFLUENZA VACCINE (SIIV) IN ADULTS ≥65 YEARS OF AGE
Brief Title: Safety and Immunogenicity of 20vPnC Coadministered With SIIV in Adults ≥65 Years of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B7471004
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Results first posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-06

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — Sodium Chloride; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Coadministration Group (Active Comparator): Participants receive injections of pneumococcal vaccine (20vPnC) and influenza vaccine at the same visit, and then receive an injection of saline 1 month later.
  Interventions: Biological: Experimental 20-valent pneumococcal conjugate vaccine (20vPnC); Other: Saline; Biological: Influenza vaccine
- Separate Administration Group (Active Comparator): Participants receive injections of saline and influenza vaccine at the same visit, and then receive an injection of 20vPnC 1 month later.
  Interventions: Biological: Experimental 20-valent pneumococcal conjugate vaccine (20vPnC); Other: Saline; Biological: Influenza vaccine

INTERVENTIONS:
Biological: Experimental 20-valent pneumococcal conjugate vaccine (20vPnC) — Experimental 20-valent pneumococcal conjugate vaccine (20vPnC)
Other: Saline — Normal saline for injection
Biological: Influenza vaccine — Seasonal inactivated influenza vaccine (SIIV)

SUMMARY:
Study of the safety and immunogenicity of 20vPnC and influenza vaccine administered at the same visit or separately

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants ≥65 years of age at the time of consent
* Adults determined by clinical assessment, including medical history and clinical judgment, to be eligible for the study, including adults with preexisting stable disease
* Adults who have no history of ever receiving a pneumococcal vaccine, or have a history of receiving a licensed pneumococcal vaccination ≥6 months prior to first study vaccination.

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis)
* Previous vaccination with any investigational pneumococcal vaccine, or planned receipt of any licensed or investigational pneumococcal vaccine through study participation.
* Vaccination with any influenza or pneumococcal vaccine <6 months before investigational product administration, or planned receipt of any licensed or investigational non-study influenza vaccine during study participation.

  -- Serious chronic disorder, that in the investigator's opinion would make the participant inappropriate for entry into the study
* Other acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1796 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (62):
- United States (62):
  - Alliance for Multispecialty Research, LLC, Mobile, Alabama
  - East Valley Gastroenterology and Hepatology Associates, Chandler, Arizona
  - Hope Research Institute, Phoenix, Arizona
  - Paradigm Clinical Research Center, Redding, California
  - Artemis Institute for Clinical Research, San Diego, California
  - California Research Foundation, San Diego, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Alliance for Multispecialty Research, LLC - Miami, Coral Gables, Florida
  - Nature Coast Clinical Research, Crystal River, Florida
  - Indago Research and Health Center, Inc., Hialeah, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - Alpha Science Research, LLC, Miami, Florida
  - Lakes Research, Miami Lakes, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Alliance for Multispecialty Research, LLC, El Dorado, Kansas
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Alliance for Multispecialty Research, LLC, New Orleans, Louisiana
  - Centennial Medical Group, Elkridge, Maryland
  - Meridian Clinical Research, LLC, Rockville, Maryland
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Meridian Clinical Research, Norfolk, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Meridian Clinical Research, LLC, Binghamton, New York
  - Meridian Clinical Research, LLC, Endwell, New York
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Accellacare - Raleigh, Raleigh, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Meridian Clinical Research, Cincinnati, Ohio
  - Velocity Clinical Research, Inc., Cleveland, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Omega Medical Research, Warwick, Rhode Island
  - Main Street Physician's Care, Little River, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Internal Medicine and Pediatric Associates of Bristol, PC, Bristol, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Benchmark Research, Austin, Texas
  - Velocity Clinical Research, Austin, Cedar Park, Texas
  - Benchmark Research, Fort Worth, Texas
  - Texas Health Resource, Fort Worth, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Wellness Clinical Research, McKinney, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - J. Lewis Research Inc. / Foothill Family Clinic Draper, Draper, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - J. Lewis Research, Inc / Jordan River Family Medicine, South Jordan, Utah
  - Alliance for Multispecialty Research - Norfolk, Norfolk, Virginia
  - National Clinical Research, Inc, Richmond, Virginia
  - Allegiance Research Specialists, LLC, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Cannon K, Cardona JF, Yacisin K, Thompson A, Belanger TJ, Lee DY, Peng Y, Moyer L, Ginis J, Gruber WC, Scott DA, Watson W. Safety and immunogenicity of a 20-valent pneumococcal conjugate vaccine coadministered with quadrivalent influenza vaccine: A phase 3 randomized trial. Vaccine. 2023 Mar 24;41(13):2137-2146. doi: 10.1016/j.vaccine.2022.11.046. Epub 2023 Feb 23. PMID 36828719
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471004

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1796 participants were enrolled in the study and assigned to a study treatment.
Groups:
- (SIIV+20vPnC)/Saline: Coadministration: On Day 1, participants received a single dose of seasonal inactivated influenza vaccine (SIIV) intramuscularly into the right deltoid along with 0.5 milliliter (mL) 20-valent pneumococcal conjugate vaccine (20vPnC) intramuscularly into the left deltoid (Vaccination 1). After one month, participants received 0.5 mL of saline intramuscularly into the left deltoid (Vaccination 2). Participants were followed up for 6 months after Vaccination 2.
- (SIIV+Saline)/20vPnC: Separate Administration: On Day 1, participants received a single dose of SIIV intramuscularly into the right deltoid and 0.5 mL of saline intramuscularly into the left deltoid (Vaccination 1). After one month, participants received 0.5 mL of 20vPnC intramuscularly into the left deltoid. (Vaccination 2). Participants were followed up for 6 months after Vaccination 2.
Period: Overall Study
Arm/Group | (SIIV+20vPnC)/Saline: Coadministration | (SIIV+Saline)/20vPnC: Separate Administration
Started | 898 | 898
Vaccination 1 | 895 | 896
Vaccination 2 | 874 | 878
Completed | 862 | 865
Not Completed | 36 | 33
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 12 | 9
Not completed — Other | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Death | 2 | 3
Not completed — Lost to Follow-up | 9 | 9
Not completed — No longer meets eligibility criteria | 8 | 8

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received 1 dose of 20vPnC or SIIV or saline and had safety follow-up after any dose.
Groups:
- (SIIV+20vPnC)/Saline: Coadministration: On Day 1, participants received a single dose of SIIV intramuscularly into the right deltoid along with 0.5 mL 20vPnC intramuscularly into the left deltoid (Vaccination 1). After one month, participants received 0.5 mL of saline intramuscularly into the left deltoid (Vaccination 2). Participants were followed up for 6 months after Vaccination 2.
- Total: Total of all reporting groups
Arm/Group | (SIIV+20vPnC)/Saline: Coadministration | (SIIV+Saline)/20vPnC: Separate Administration | Total
Number analyzed (Participants) | 895 | 896 | 1791
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.1 (5.49) | 71.9 (5.48) | 72.0 (5.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 483 | 496 | 979
  Male | 412 | 400 | 812
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 92 | 77 | 169
  Not Hispanic or Latino | 793 | 813 | 1606
  Unknown or Not Reported | 10 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 7 | 15 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 58 | 65 | 123
  White | 816 | 807 | 1623
  More than one race | 10 | 3 | 13
  Unknown or Not Reported | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 10 Days After Vaccination With 20vPnC
Description: Local reactions were collected at the 20vPnC injection sites after Vaccination 1 and Vaccination 2 and were recorded by the participants using an electronic diary (e-diary). Local reactions included redness, swelling and pain at the injection site. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm). Redness and swelling were graded as mild (greater than [>] 2.0 to 5.0 cm), moderate (>5.0 to 10.0 cm) and severe (>10.0 cm). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), and severe (prevented daily activity). Percentage of participants with local reactions at the 20vPnC injection site in the Coadministration group and the Separate administration group and the associated 2-sided 95% confidence interval (CI) based on the Clopper and Pearson method was presented.
Time Frame: Within 10 days after Vaccination 1 for Coadministration group and within 10 days after Vaccination 2 for Separate Administration group
Population: Safety population included all randomized participants who received 1 dose of 20vPnC or SIIV or saline and had safety follow-up after any dose. Here, "Overall Number of Participants Analyzed" (N) signifies number of participants with any e-diary data reported after vaccination with 20vPnC.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | (SIIV+20vPnC)/Saline: Coadministration | (SIIV+Saline)/20vPnC: Separate Administration
Number analyzed (Participants) | 876 | 855
Percentage of participants
  Redness: Any | 6.3 [4.8 to 8.1] | 7.4 [5.7 to 9.3]
  Redness: Mild | 4.0 [2.8 to 5.5] | 3.3 [2.2 to 4.7]
  Redness: Moderate | 2.1 [1.2 to 3.2] | 3.3 [2.2 to 4.7]
  Redness: Severe | 0.2 [0.0 to 0.8] | 0.8 [0.3 to 1.7]
  Swelling: Any | 8.2 [6.5 to 10.2] | 7.8 [6.1 to 9.8]
  Swelling: Mild | 5.0 [3.7 to 6.7] | 4.4 [3.2 to 6.0]
  Swelling: Moderate | 2.9 [1.9 to 4.2] | 3.3 [2.2 to 4.7]
  Swelling: Severe | 0.3 [0.1 to 1.0] | 0.1 [0.0 to 0.6]
  Pain at the injection site: Any | 48.9 [45.5 to 52.2] | 51.5 [48.1 to 54.9]
  Pain at the injection site: Mild | 41.0 [37.7 to 44.3] | 42.9 [39.6 to 46.3]
  Pain at the injection site: Moderate | 7.6 [6.0 to 9.6] | 8.4 [6.6 to 10.5]
  Pain at the injection site: Severe | 0.2 [0.0 to 0.8] | 0.1 [0.0 to 0.6]

2. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Each Vaccination By Each Vaccine
Description: Systemic events including fever, fatigue, headache, muscle pain and joint pain were recorded by participants using an e-diary. Fever was defined as temperature >=38.0 degree Celsius (C) and categorized as >=38.0 to 38.4 degree C, >38.4 to 38.9 degree C, >38.9 to 40.0 degree C and >40.0 degree C. Fatigue, headache, muscle pain and joint pain were graded as mild (did not interfere with activity), moderate (some interference with activity) and severe (prevented daily routine activity). Percentage of participants with systemic events within 7 days after each vaccination and the associated 2-sided 95% CI based on the Clopper and Pearson method was presented.
Time Frame: Within 7 days after each vaccination
Population: Safety population included all randomized participants who received 1 dose of 20vPnC or SIIV or saline and had safety follow-up after any dose. Here, 'N' signifies number of participants with any e-diary data reported after the vaccination at the specified visit.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- 20vPnC Coadministered With SIIV: Participants in the (SIIV+20vPnC)/Saline (Coadministration) group received a single dose of SIIV intramuscularly into the right deltoid along with 0.5 mL 20vPnC intramuscularly into the left deltoid (Vaccination 1).
- Separate SIIV Administration: Participants in the (SIIV+Saline)/20vPnC group received single dose of SIIV injected intramuscularly into the left deltoid (Vaccination 1).
- Saline Only: Participants in the (SIIV+20vPnC)/Saline: Coadministration group received 0.5 mL of saline intramuscularly into the left deltoid (Vaccination 2), one month after Vaccination 1.
- Separate 20vPnC: Participants in the (SIIV+Saline)/20vPnC group received single dose of 0.5 ml of 20vPnC injected intramuscularly into the left deltoid (Vaccination 2), one month after Vaccination 1.
Arm/Group | 20vPnC Coadministered With SIIV | Separate SIIV Administration | Saline Only | Separate 20vPnC
Number analyzed (Participants) | 877 | 883 | 853 | 855
Percentage of participants
  Fever: >=38.0 degree C | 1.5 [0.8 to 2.5] | 0.6 [0.2 to 1.3] | 0.7 [0.3 to 1.5] | 0.5 [0.1 to 1.2]
  Fever: >=38.0 degree C to 38.4 degree C | 0.9 [0.4 to 1.8] | 0.5 [0.1 to 1.2] | 0.6 [0.2 to 1.4] | 0.4 [0.1 to 1.0]
  Fever: >38.4 degree C to 38.9 degree C | 0.5 [0.1 to 1.2] | 0.1 [0.0 to 0.6] | 0 [0.0 to 0.4] | 0.1 [0.0 to 0.6]
  Fever: >38.9 degree C to 40.0 degree C | 0.1 [0.0 to 0.6] | 0 [0.0 to 0.4] | 0.1 [0.0 to 0.7] | 0 [0.0 to 0.4]
  Fever: >40.0 degree C | 0 [0.0 to 0.4] | 0 [0.0 to 0.4] | 0 [0.0 to 0.4] | 0 [0.0 to 0.4]
  Fatigue: Any | 33.2 [30.1 to 36.4] | 22.8 [20.0 to 25.7] | 13.2 [11.0 to 15.7] | 20.1 [17.5 to 23.0]
  Fatigue: Mild | 20.0 [17.4 to 22.8] | 12.6 [10.5 to 14.9] | 8.0 [6.2 to 10.0] | 10.8 [8.8 to 13.0]
  Fatigue: Moderate | 12.3 [10.2 to 14.7] | 9.6 [7.8 to 11.8] | 4.9 [3.6 to 6.6] | 8.4 [6.6 to 10.5]
  Fatigue: Severe | 0.9 [0.4 to 1.8] | 0.6 [0.2 to 1.3] | 0.4 [0.1 to 1.0] | 0.9 [0.4 to 1.8]
  Headache: Any | 21.9 [19.2 to 24.8] | 18.0 [15.5 to 20.7] | 12.0 [9.9 to 14.3] | 15.3 [13.0 to 17.9]
  Headache: Mild | 16.2 [13.8 to 18.8] | 13.0 [10.9 to 15.4] | 9.1 [7.3 to 11.3] | 10.9 [8.9 to 13.2]
  Headache: Moderate | 5.5 [4.1 to 7.2] | 5.0 [3.6 to 6.6] | 2.6 [1.6 to 3.9] | 4.1 [2.9 to 5.6]
  Headache: Severe | 0.2 [0.0 to 0.8] | 0 [0.0 to 0.4] | 0.2 [0.0 to 0.8] | 0.4 [0.1 to 1.0]
  Muscle Pain: Any | 19.7 [17.1 to 22.5] | 13.7 [11.5 to 16.1] | 8.2 [6.5 to 10.3] | 14.2 [11.9 to 16.7]
  Muscle Pain: Mild | 11.1 [9.1 to 13.3] | 8.9 [7.1 to 11.0] | 4.2 [3.0 to 5.8] | 8.8 [7.0 to 10.9]
  Muscle Pain: Moderate | 8.0 [6.3 to 10.0] | 4.5 [3.3 to 6.1] | 3.9 [2.7 to 5.4] | 5.4 [4.0 to 7.1]
  Muscle Pain: Severe | 0.7 [0.3 to 1.5] | 0.2 [0.0 to 0.8] | 0.1 [0.0 to 0.7] | 0 [0.0 to 0.4]
  Joint Pain: Any | 13.3 [11.2 to 15.8] | 12.5 [10.4 to 14.8] | 7.7 [6.0 to 9.7] | 10.3 [8.3 to 12.5]
  Joint Pain: Mild | 6.6 [5.1 to 8.5] | 6.6 [5.0 to 8.4] | 2.7 [1.7 to 4.0] | 6.4 [4.9 to 8.3]
  Joint Pain: Moderate | 6.5 [5.0 to 8.3] | 5.7 [4.2 to 7.4] | 4.8 [3.5 to 6.5] | 3.6 [2.5 to 5.1]
  Joint Pain: Severe | 0.2 [0.0 to 0.8] | 0.2 [0.0 to 0.8] | 0.2 [0.0 to 0.8] | 0.2 [0.0 to 0.8]

3. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Each Vaccination by Each Vaccine
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Within 1 month after each vaccination
Population: Safety population included all randomized participants who received 1 dose of 20vPnC or SIIV or saline and had safety follow-up after any dose. Here, 'Overall number of participants analyzed' (N) is the number of participants included in the safety population who received the specified vaccination.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 20vPnC Coadministered With SIIV | Separate SIIV Administration | Saline Only | Separate 20vPnC
Number analyzed (Participants) | 895 | 896 | 874 | 878
Percentage of participants | 9.1 [7.3 to 11.1] | 8.0 [6.3 to 10.0] | 6.3 [4.8 to 8.1] | 8.7 [6.9 to 10.7]

4. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) From the First Vaccination up to 6 Months After Last Vaccination
Description: An SAE was defined as any untoward medical occurrence that, at any dose that results in death; is life-threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect or that is considered to be an important medical event. Percentage of participants with SAEs and the associated 2-sided 95% CI based on the Clopper and Pearson method was presented.
Time Frame: From Day 1 up to 6 months after last Vaccination (i.e. up to 7 months)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | (SIIV+20vPnC)/Saline: Coadministration | (SIIV+Saline)/20vPnC: Separate Administration
Number analyzed (Participants) | 895 | 896
Percentage of participants | 3.7 [2.6 to 5.1] | 3.7 [2.5 to 5.1]

5. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Condition (NDCMC) up to 6 Months After Last Vaccination
Description: An NDCMC was defined as a significant disease or medical condition, not previously identified, that is expected to be persistent or is otherwise long-lasting in its effects. Percentage of participants with NDCMC and the associated 2-sided 95% CI based on the Clopper and Pearson method was presented.
Time Frame: Up to 6 months after last Vaccination (i.e. up to 7 months)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | (SIIV+20vPnC)/Saline: Coadministration | (SIIV+Saline)/20vPnC: Separate Administration
Number analyzed (Participants) | 895 | 896
Percentage of participants | 3.8 [2.6 to 5.3] | 3.1 [2.1 to 4.5]

6. Primary Outcome: Model-Based Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) at 1 Month After Vaccination With 20vPnC
Description: OPA titers were measured from serum samples for 20vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F,8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, 33F. GMTs and 2-sided CIs were calculated by exponentiating the LS means and the corresponding CIs based on analysis of log-transformed OPA titers using a regression model
Time Frame: 1 month after the 20vPnC administration in each group (1 month after Vaccination 1 in the Coadministration group and 1 month after Vaccination 2 in the Separate Administration group).
Population: Evaluable pneumococcal immunogenicity(EPI) population: all randomized participants who received assigned vaccinations; blood collected within 27 to 49 days after 20vPnC; with least 1 valid OPA result from sample collected 1 month after 20vPnC vaccination; had no other major protocol deviations as determined by clinician. Here,'N':number of participants in evaluable immunogenicity population and 'number analyzed': number of evaluable participants with a valid OPA titer for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | (SIIV+20vPnC)/Saline: Coadministration | (SIIV+Saline)/20vPnC: Separate Administration
Number analyzed (Participants) | 854 | 834
Titer
  Serotype 1: number analyzed (Participants) | 851 | 830
  Serotype 1 | 70 [63 to 79] | 95 [85 to 107]
  Serotype 3: number analyzed (Participants) | 846 | 828
  Serotype 3 | 38 [34 to 41] | 46 [42 to 50]
  Serotype 4: number analyzed (Participants) | 838 | 828
  Serotype 4 | 567 [500 to 642] | 639 [563 to 724]
  Serotype 5: number analyzed (Participants) | 850 | 824
  Serotype 5 | 71 [64 to 78] | 81 [73 to 89]
  Serotype 6A: number analyzed (Participants) | 838 | 825
  Serotype 6A | 753 [657 to 863] | 995 [868 to 1141]
  Serotype 6B: number analyzed (Participants) | 844 | 823
  Serotype 6B | 855 [754 to 971] | 1050 [923 to 1194]
  Serotype 7F: number analyzed (Participants) | 848 | 830
  Serotype 7F | 918 [846 to 996] | 1015 [936 to 1101]
  Serotype 8: number analyzed (Participants) | 823 | 814
  Serotype 8 | 260 [228 to 296] | 323 [284 to 368]
  Serotype 9V: number analyzed (Participants) | 829 | 823
  Serotype 9V | 1261 [1115 to 1426] | 1344 [1189 to 1519]
  Serotype 10A: number analyzed (Participants) | 804 | 793
  Serotype 10A | 1391 [1213 to 1595] | 1681 [1468 to 1925]
  Serotype 11A: number analyzed (Participants) | 793 | 773
  Serotype 11A | 1032 [886 to 1202] | 1453 [1249 to 1690]
  Serotype 12F: number analyzed (Participants) | 814 | 779
  Serotype 12F | 1352 [1161 to 1574] | 1652 [1415 to 1929]
  Serotype 14: number analyzed (Participants) | 845 | 823
  Serotype 14 | 514 [463 to 571] | 600 [540 to 667]
  Serotype 15B: number analyzed (Participants) | 800 | 779
  Serotype 15B | 839 [695 to 1012] | 1202 [997 to 1450]
  Serotype 18C: number analyzed (Participants) | 846 | 828
  Serotype 18C | 825 [723 to 943] | 920 [805 to 1051]
  Serotype 19A: number analyzed (Participants) | 845 | 831
  Serotype 19A | 467 [420 to 519] | 534 [480 to 593]
  Serotype 19F: number analyzed (Participants) | 847 | 822
  Serotype 19F | 241 [215 to 270] | 272 [243 to 305]
  Serotype 22F: number analyzed (Participants) | 771 | 774
  Serotype 22F | 2192 [1850 to 2597] | 2933 [2481 to 3468]
  Serotype 23F: number analyzed (Participants) | 849 | 831
  Serotype 23F | 247 [213 to 287] | 318 [273 to 369]
  Serotype 33F: number analyzed (Participants) | 800 | 791
  Serotype 33F | 3047 [2672 to 3475] | 4259 [3737 to 4853]
Statistical Analysis 1: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 1: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of least square (LS) means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — Noninferiority (NI) for a serotype was declared if the lower bound of the 2-sided 95% CI for the GMR of the (SIIV+20vPnC)/saline group to the (SIIV+saline)/20vPnC group was greater than 0.5 (2-fold criterion) for that serotype; Geometric Mean Ratio (GMR) = 0.74, 95% CI 2-sided [0.65 to 0.84]
Statistical Analysis 2: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 3: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — NI for a serotype was declared if the lower bound of the 2-sided 95% CI for the GMR of the (SIIV+20vPnC)/saline group to the (SIIV+saline)/20vPnC group was greater than 0.5 (2-fold criterion) for that serotype; GMR = 0.82, 95% CI 2-sided [0.75 to 0.90]
Statistical Analysis 3: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 4: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.89, 95% CI 2-sided [0.77 to 1.02]
Statistical Analysis 4: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 5: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.88, 95% CI 2-sided [0.79 to 0.98]
Statistical Analysis 5: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 6A: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.76, 95% CI 2-sided [0.65 to 0.88]
Statistical Analysis 6: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 6B: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.81, 95% CI 2-sided [0.71 to 0.94]
Statistical Analysis 7: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 7F: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.90, 95% CI 2-sided [0.83 to 0.99]
Statistical Analysis 8: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 8: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.80, 95% CI 2-sided [0.70 to 0.93]
Statistical Analysis 9: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 9V: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.94, 95% CI 2-sided [0.82 to 1.07]
Statistical Analysis 10: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 10A: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.83, 95% CI 2-sided [0.71 to 0.96]
Statistical Analysis 11: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 11A: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.71, 95% CI 2-sided [0.60 to 0.84]
Statistical Analysis 12: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 12F: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.82, 95% CI 2-sided [0.69 to 0.97]
Statistical Analysis 13: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 14: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.86, 95% CI 2-sided [0.76 to 0.96]
Statistical Analysis 14: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 15B: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.70, 95% CI 2-sided [0.57 to 0.86]
Statistical Analysis 15: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 18C: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.90, 95% CI 2-sided [0.77 to 1.04]
Statistical Analysis 16: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 19A: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.88, 95% CI 2-sided [0.78 to 0.98]
Statistical Analysis 17: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 19F: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.89, 95% CI 2-sided [0.78 to 1.01]
Statistical Analysis 18: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 22F: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.75, 95% CI 2-sided [0.62 to 0.90]
Statistical Analysis 19: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 23F: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.78, 95% CI 2-sided [0.66 to 0.92]
Statistical Analysis 20: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; Serotype 33F: GMR (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 95% CIs were calculated by exponentiating the difference of LS means for OPA titers and corresponding CIs based on regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed OPA titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 2]; GMR = 0.72, 95% CI 2-sided [0.62 to 0.83]

7. Primary Outcome: Model-Based Hemagglutination Inhibition (HAI) Strain Specific Geometric Mean Titers (GMT) at 1 Month After Vaccination With SIIV
Description: HAI titers to the influenza strains (A/H1N1, A/H3N2, B/Victoria, and B/Phuket) in the SIIV administered sera samples was collected and reported in this outcome measure at 1 month after Vaccination 1. GMTs and 2-sided CIs were calculated by exponentiating the LS means and the corresponding CIs based on analysis of log-transformed HAI titers using a regression model.
Time Frame: At 1 month after Vaccination 1 with SIIV
Population: Evaluable HAI immunogenicity population: all randomized participants who received assigned vaccinations; had blood collected within 27 to 49 days after SIIV; had at least 1 valid HAI result from blood sample collected 1 month after SIIV vaccination; had no other major protocol deviations as determined by clinician. Here, 'N': number of participants in evaluable HAI immunogenicity population, 'number analyzed': number of evaluable HAI participants with a valid result for the specified HAI strain.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | (SIIV+20vPnC)/Saline: Coadministration | (SIIV+Saline)/20vPnC: Separate Administration
Number analyzed (Participants) | 861 | 865
Titer
  A/H1N1 | 51.9 [47.6 to 56.6] | 48.7 [44.7 to 53.0]
  A/H3N2 | 189.8 [173.9 to 207.2] | 193.4 [177.3 to 211.0]
  B/Victoria | 68.1 [63.4 to 73.1] | 68.0 [63.4 to 73.0]
  B/Phuket | 39.4 [36.3 to 42.6] | 41.6 [38.4 to 45.0]
Statistical Analysis 1: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; A/H1N1: GMRs (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 2-sided CIs were calculated by exponentiating the difference of LS means for the HAI titers and the corresponding CIs based on the regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed HAI titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — NI was declared if the lower bound of the 2-sided 95% CI for the GMR of the (SIIV+20vPnC)/saline group to the (SIIV+saline)/20vPnC group was greater than 0.67 (1.5-fold criterion); GMR = 1.07, 95% CI 2-sided [0.97 to 1.17]
Statistical Analysis 2: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; A/H3N2: GMRs (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 2-sided CIs were calculated by exponentiating the difference of LS means for the HAI titers and the corresponding CIs based on the regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed HAI titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; GMR = 0.98, 95% CI 2-sided [0.89 to 1.08]
Statistical Analysis 3: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; B/Victoria: GMRs (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 2-sided CIs were calculated by exponentiating the difference of LS means for the HAI titers and the corresponding CIs based on the regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed HAI titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; GMR = 1.00, 95% CI 2-sided [0.93 to 1.08]
Statistical Analysis 4: Comparison: (SIIV+20vPnC)/Saline: Coadministration vs (SIIV+Saline)/20vPnC: Separate Administration; B/Phuket: GMRs (ratio of GMTs [SIIV+20vPnC]/saline to [SIIV+saline]/20vPnC) and 2-sided CIs were calculated by exponentiating the difference of LS means for the HAI titers and the corresponding CIs based on the regression model adjusted with vaccine group, sex, smoking status, age at Vaccination 1 in years, baseline log-transformed HAI titers, and prior pneumococcal vaccination status; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; GMR = 0.95, 95% CI 2-sided [0.87 to 1.03]

8. Secondary Outcome: Percentage of Participants With Greater Than or Equal to (≥4) Fold Rise in Serotype-Specific Opsonophagocytic Activity (OPA) Titers From Before Vaccination to 1 Month After Vaccination With 20vPnC
Description: OPA titers were measured from serum samples for 20vPnC serotypes: 1, 3, 4, 5, 6A, 6B, 7F,8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, 33F. Percentage of participants with >=4 fold rise in serotype-specific OPA titers from before vaccination to 1 month after vaccination with 20vPnC and the associated 2-sided 95% CI based on the Clopper and Pearson method was presented.
Time Frame: Before Vaccination 1 to 1 month after 20vPnC vaccination in both groups (i.e., 1 month after Vaccination 1 in Coadministration group and 1 month after Vaccination 2 in Separate Administration group)
Population: EPI population: all randomized participants who received assigned vaccinations; blood collected within 27 to 49 days after 20vPnC with at least 1 valid OPA result from sample collected 1 month after 20vPnC vaccination; no other major protocol deviations as determined by clinician. Here, 'N': number of participants with valid results for both timepoints (before Vaccination 1 and 1 month after 20vPnC), 'number analyzed': participants evaluable for specific serotypes.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | (SIIV+20vPnC)/Saline: Coadministration | (SIIV+Saline)/20vPnC: Separate Administration
Number analyzed (Participants) | 854 | 834
Percentage of participants
  Serotype 1: number analyzed (Participants) | 845 | 824
  Serotype 1 | 32.9 [29.7 to 36.2] | 42.0 [38.6 to 45.4]
  Serotype 3: number analyzed (Participants) | 836 | 819
  Serotype 3 | 31.1 [28.0 to 34.4] | 39.7 [36.3 to 43.1]
  Serotype 4: number analyzed (Participants) | 814 | 796
  Serotype 4 | 45.3 [41.9 to 48.8] | 48.5 [45.0 to 52.0]
  Serotype 5: number analyzed (Participants) | 844 | 817
  Serotype 5 | 28.2 [25.2 to 31.4] | 32.7 [29.5 to 36.0]
  Serotype 6A: number analyzed (Participants) | 818 | 800
  Serotype 6A | 57.7 [54.2 to 61.1] | 62.9 [59.4 to 66.2]
  Serotype 6B: number analyzed (Participants) | 826 | 801
  Serotype 6B | 51.7 [48.2 to 55.2] | 55.3 [51.8 to 58.8]
  Serotype 7F: number analyzed (Participants) | 820 | 806
  Serotype 7F | 26.5 [23.5 to 29.6] | 29.3 [26.2 to 32.6]
  Serotype 8: number analyzed (Participants) | 797 | 785
  Serotype 8 | 52.1 [48.5 to 55.6] | 53.8 [50.2 to 57.3]
  Serotype 9V: number analyzed (Participants) | 797 | 789
  Serotype 9V | 41.4 [38.0 to 44.9] | 43.6 [40.1 to 47.1]
  Serotype 10A: number analyzed (Participants) | 757 | 755
  Serotype 10A | 56.5 [52.9 to 60.1] | 62.0 [58.4 to 65.5]
  Serotype 11A: number analyzed (Participants) | 708 | 690
  Serotype 11A | 43.5 [39.8 to 47.2] | 50.6 [46.8 to 54.4]
  Serotype 12F: number analyzed (Participants) | 782 | 741
  Serotype 12F | 60.1 [56.6 to 63.6] | 63.6 [60.0 to 67.0]
  Serotype 14: number analyzed (Participants) | 824 | 808
  Serotype 14 | 24.8 [21.8 to 27.9] | 30.3 [27.2 to 33.6]
  Serotype 15B: number analyzed (Participants) | 758 | 750
  Serotype 15B | 56.7 [53.1 to 60.3] | 60.8 [57.2 to 64.3]
  Serotype 18C: number analyzed (Participants) | 833 | 818
  Serotype 18C | 39.3 [35.9 to 42.7] | 42.7 [39.2 to 46.1]
  Serotype 19A: number analyzed (Participants) | 827 | 816
  Serotype 19A | 36.0 [32.8 to 39.4] | 40.2 [36.8 to 43.7]
  Serotype 19F: number analyzed (Participants) | 841 | 810
  Serotype 19F | 33.9 [30.7 to 37.2] | 38.6 [35.3 to 42.1]
  Serotype 22F: number analyzed (Participants) | 699 | 707
  Serotype 22F | 68.7 [65.1 to 72.1] | 72.0 [68.5 to 75.3]
  Serotype 23F: number analyzed (Participants) | 840 | 822
  Serotype 23F | 49.8 [46.3 to 53.2] | 55.1 [51.6 to 58.5]
  Serotype 33F: number analyzed (Participants) | 760 | 750
  Serotype 33F | 39.1 [35.6 to 42.7] | 47.7 [44.1 to 51.4]

9. Secondary Outcome: Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rise (GMFR) From Before Vaccination to 1 Month After Vaccination With 20vPnC
Description: OPA titers were measured from serum samples for serotypes: 1, 3, 4, 5, 6A, 6B, 7F,8, 9V, 10A, 11A, 12F, 14, 15B, 18C, 19A, 19F, 22F, 23F, 33F. GMFR was calculated as geometric mean of fold rise from before vaccination on Day 1 to 1 month after vaccination with 20vPnC. GMFRs and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the OPA titers or fold rises and the corresponding CIs.
Time Frame: as for outcome 8
Population: EPI population: all randomized participants who received assigned vaccinations; blood collected within 27 to 49 days after 20vPnC with at least 1 valid OPA result from sample collected 1 month after 20vPnC vaccination; no other major protocol deviations as determined by clinician. Here, 'N': number of participants in the EPI, 'number analyzed': participants with valid OPA titers both before vaccination at Visit 1 and 1 month after 20vPnC blood sample collections.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | (SIIV+20vPnC)/Saline: Coadministration | (SIIV+Saline)/20vPnC: Separate Administration
Number analyzed (Participants) | 854 | 834
Fold rise
  Serotype 1: number analyzed (Participants) | 845 | 824
  Serotype 1 | 3.0 [2.8 to 3.3] | 4.0 [3.6 to 4.5]
  Serotype 3: number analyzed (Participants) | 836 | 819
  Serotype 3 | 2.5 [2.3 to 2.7] | 3.1 [2.8 to 3.3]
  Serotype 4: number analyzed (Participants) | 814 | 796
  Serotype 4 | 6.2 [5.4 to 7.1] | 7.4 [6.4 to 8.5]
  Serotype 5: number analyzed (Participants) | 844 | 817
  Serotype 5 | 2.4 [2.2 to 2.6] | 2.7 [2.5 to 3.0]
  Serotype 6A: number analyzed (Participants) | 818 | 800
  Serotype 6A | 8.8 [7.7 to 10.1] | 11.9 [10.4 to 13.7]
  Serotype 6B: number analyzed (Participants) | 826 | 801
  Serotype 6B | 6.5 [5.8 to 7.3] | 8.4 [7.4 to 9.5]
  Serotype 7F: number analyzed (Participants) | 820 | 806
  Serotype 7F | 2.6 [2.4 to 2.8] | 2.8 [2.5 to 3.1]
  Serotype 8: number analyzed (Participants) | 797 | 785
  Serotype 8 | 5.8 [5.1 to 6.6] | 7.3 [6.3 to 8.3]
  Serotype 9V: number analyzed (Participants) | 797 | 789
  Serotype 9V | 4.0 [3.6 to 4.5] | 4.3 [3.8 to 4.8]
  Serotype 10A: number analyzed (Participants) | 757 | 755
  Serotype 10A | 8.0 [7.0 to 9.2] | 10.1 [8.8 to 11.6]
  Serotype 11A: number analyzed (Participants) | 708 | 690
  Serotype 11A | 4.4 [3.9 to 5.1] | 6.2 [5.3 to 7.1]
  Serotype 12F: number analyzed (Participants) | 782 | 741
  Serotype 12F | 11.4 [9.7 to 13.3] | 14.4 [12.2 to 17.0]
  Serotype 14: number analyzed (Participants) | 824 | 808
  Serotype 14 | 2.5 [2.3 to 2.8] | 3.0 [2.7 to 3.4]
  Serotype 15B: number analyzed (Participants) | 758 | 750
  Serotype 15B | 11.7 [9.9 to 14.0] | 16.4 [13.6 to 19.8]
  Serotype 18C: number analyzed (Participants) | 833 | 818
  Serotype 18C | 4.6 [4.0 to 5.2] | 5.2 [4.5 to 5.9]
  Serotype 19A: number analyzed (Participants) | 827 | 816
  Serotype 19A | 3.7 [3.3 to 4.1] | 4.2 [3.8 to 4.7]
  Serotype 19F: number analyzed (Participants) | 841 | 810
  Serotype 19F | 3.0 [2.7 to 3.3] | 3.3 [3.0 to 3.7]
  Serotype 22F: number analyzed (Participants) | 699 | 707
  Serotype 22F | 23.6 [19.4 to 28.6] | 32.3 [26.5 to 39.4]
  Serotype 23F: number analyzed (Participants) | 840 | 822
  Serotype 23F | 6.4 [5.6 to 7.2] | 8.5 [7.4 to 9.7]
  Serotype 33F: number analyzed (Participants) | 760 | 750
  Serotype 33F | 3.3 [3.0 to 3.7] | 4.8 [4.2 to 5.4]

10. Secondary Outcome: Hemagglutination Inhibition (HAI) Strain Specific Geometric Mean Fold Rise (GMFR) Before Vaccination to 1 Month After Vaccination With SIIV
Description: HAI titers were measured from serum samples for serotypes A/H1N1, A/H3N2, B/Victoria, B/Phuket. GMFR was calculated as geometric mean of fold rise from before vaccination on Day 1 to 1 month after vaccination with SIIV. GMFRs were calculated for participants with non-missing values both before and after vaccination.
Time Frame: Before Vaccination 1 to 1 month after Vaccination 1 with SIIV
Population: Evaluable HAI immunogenicity population:randomized participants who received assigned vaccinations; blood collected within 27 to 49 days after SIIV;had at least 1 valid HAI result from blood sample collected 1 month after SIIV vaccination; no other major protocol deviations as determined by clinician. 'N': participants analyzed in HAI immunogenicity population, 'number analyzed':participants with valid HAI titers both before vaccination at Visit 1 and 1 month after SIIV blood sample collections.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | (SIIV+20vPnC)/Saline: Coadministration | (SIIV+Saline)/20vPnC: Separate Administration
Number analyzed (Participants) | 861 | 865
Fold rise
  A/H1N1: number analyzed (Participants) | 860 | 864
  A/H1N1 | 1.8 [1.7 to 2.0] | 1.8 [1.6 to 2.0]
  A/H3N2: number analyzed (Participants) | 860 | 864
  A/H3N2 | 2.0 [1.8 to 2.2] | 2.0 [1.8 to 2.2]
  B/Victoria: number analyzed (Participants) | 860 | 864
  B/Victoria | 1.7 [1.6 to 1.8] | 1.7 [1.6 to 1.9]
  B/Phuket: number analyzed (Participants) | 860 | 864
  B/Phuket | 1.4 [1.3 to 1.5] | 1.4 [1.3 to 1.5]

ADVERSE EVENTS:
Time Frame: Local reactions(systematic assessment): within 10 days after Vaccination 1 for Coadministration group and within 10 days after Vaccination 2 for Separate Administration group, Systemic events(systematic assessment): within 7 days after Vaccination 1 for Coadministration group and within 7 days after Vaccination 2 for Separate Administration group, SAEs: from Day 1 up to 6 months after last vaccination(i.e., up to 7 months) and other AEs: up to 1 month after each vaccination
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study.
Arm/Group | (SIIV+20vPnC)/Saline: Coadministration | (SIIV+Saline)/20vPnC: Separate Administration
All-Cause Mortality (participants affected / at risk) | 2/895 | 3/896
Serious Adverse Events (participants affected / at risk) | 33/895 | 33/896
Other Adverse Events (participants affected / at risk) | 629/895 | 644/896
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | (SIIV+20vPnC)/Saline: Coadministration (N=895) | (SIIV+Saline)/20vPnC: Separate Administration (N=896)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrioventricular block complete (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 2 | 2
Vascular stent stenosis (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 3
COVID-19 pneumonia (Infections and infestations) | 3 | 1
Cellulitis (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | (SIIV+20vPnC)/Saline: Coadministration (N=895) | (SIIV+Saline)/20vPnC: Separate Administration (N=896)
Fatigue (FATIGUE) (General disorders) | 332 | 299
Injection site erythema (REDNESS) (General disorders) | 57 | 67
Injection site pain (PAIN) (General disorders) | 440 | 461
Injection site swelling (SWELLING) (General disorders) | 73 | 76
Pyrexia (FEVER) (General disorders) | 17 | 9
COVID-19 (Infections and infestations) | 12 | 18
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 148 | 155
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 207 | 199
Headache (HEADACHE) (Nervous system disorders) | 241 | 231
Fall (Injury, poisoning and procedural complications) | 11 | 12
SARS-CoV-2 test positive (Investigations) | 14 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT04526574/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT04526574/SAP_001.pdf